CLINICAL TRIAL: NCT04960033
Title: Central South University
Brief Title: Evaluating Fracture Risk Assessment Tools (FRAX) From Different Regions in Central South Chinese Postmenopausal Women
Status: Completed | Type: Observational
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, ChenRong, Central South University, Central South University
Other Study IDs: Sheng zhifeng
Record Dates: First submitted 2021-07-02; First posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Osteoporosis Fracture
Keywords: FRAX; osteoporosis; Chinese population
MeSH Terms: conditions — Osteoporotic Fractures; Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Osteoporosis fracture: The 10-year MOF probability and the 10-year HF probability were calculated using the FRAXs of different regions (mainland China, Hong Kong, Taiwan, and Asia-America). Subjects were deemed as high-risk for osteoporotic fracture if the 10-year probability of MOF was ≥20% or the 10-year probability of HF was ≥3%.
  Interventions: Behavioral: FRAX
- women without osteoporosis fracture: The 10-year MOF probability and the 10-year HF probability were calculated using the FRAXs of different regions (mainland China, Hong Kong, Taiwan, and Asia-America). Subjects were deemed as high-risk for osteoporotic fracture if the 10-year probability of MOF was <20% or the 10-year probability of HF was <3%.
  Interventions: Behavioral: FRAX

INTERVENTIONS:
Behavioral: FRAX — The 10-year MOF probability and the 10-year HF probability were calculated using the FRAXs of different regions (mainland China, Hong Kong, Taiwan, and Asia-America). Subjects were deemed as high-risk for osteoporotic fracture if the 10-year probability of MOF was ≥20% or the 10-year probability of HF was ≥3%.

SUMMARY:
We evaluated fracture risk assessment tools (FRAXs) from different regions in Chinese postmenopausal women.

DETAILED DESCRIPTION:
This cross-sectional study recruited 264 postmenopausal women aged ≥50 years in September 2017. Basic information, general condition, history of illness, family history, and clinical risk factors were evaluated via a questionnaire. All subjects underwent a bone mineral density examination of the femur and lumbar spine and thoracolumbar spinal X-ray. The 10-year major osteoporotic fracture (MOF) and hip fracture (HF) risks were calculated using FRAXs from mainland China, Hong Kong, Taiwan, and Asia-America. All data were analyzed using SPSS 17.0. Sensitivity, specificity, and likelihood ratio were used to compare the effectiveness of each FRAX.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women aged ≥50 years were randomly selected from community centers in Changsha City, Hunan Province, China in September 2017. Menopause was defined as the absence of menstrual cycles for at least one year. All subjects were noninstitutionalized and in good health.

Exclusion Criteria:

* The criteria for exclusion were morphological abnormalities or skeletal distortions that prohibited either clinical measurements or morphometric assessments of skeletal radiographs.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women aged ≥50 years were randomly selected from community centers in Changsha City, Hunan Province, China in September 2017.
Sampling Method: Probability Sample
Enrollment: 264 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Osteoporosis fracture | 2017years
  The 10-year MOF probability and the 10-year HF probability were calculated using the FRAXs of different regions (mainland China, Hong Kong, Taiwan, and Asia-America). Subjects were deemed as high-risk for osteoporotic fracture if the 10-year probability of MOF was ≥20% or the 10-year probability of HF was ≥3%.

CONTACTS AND LOCATIONS:
Locations (1):
- The 2nd Xiangya Hospital, Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhang Z, Ou Y, Sheng Z, Liao E. How to decide intervention thresholds based on FRAX in central south Chinese postmenopausal women. Endocrine. 2014 Mar;45(2):195-7. doi: 10.1007/s12020-013-0076-y. Epub 2013 Oct 22. PMID 24146412